CLINICAL TRIAL: NCT02873624
Title: Incidence of Acute Kidney Injury After Laparoscopic Cholecystectomy
Status: Terminated | Type: Observational
Why Stopped: No patients recruited
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Khaled Khazim, MD, Nephrology specialist, Western Galilee Hospital-Nahariya
Other Study IDs: WGH160112ctil
Record Dates: First submitted 2016-08-11; First posted 2016-08-19 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Acute Kidney Injury ,Laparoscopic Cholecystectomy
Keywords: Acute Kidney Injury , Laparoscopic Cholecystectomy
MeSH Terms: conditions — Acute Kidney Injury | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy

SUMMARY:
The aim of this study is to establish AKI incidence in patients who are undergoing laparoscopic cholecystectomy and to identify the potential risk factors associated with the development of AKI.

DETAILED DESCRIPTION:
Introduction: Laparoscopic procedure produces adverse effects on splanchnic organs. Pneumoperitoneum is a non-physiologic condition that causes a higher intra-abdominal pressure (IAP) and is associated with significant direct and indirect effects on renal physiology.

Aim of the study:

To establish AKI incidence in patients who are undergoing laparoscopic cholecystectomy.

To identify the potential risk factors associated with the development of AKI. To establish the relationship between the IAP during the procedure and the AKI incidence.

Study Design:

Study population: A single center prospective cohort study will be conducted. 100 patients undergoing elective laparoscopic cholecystectomy in the Galilee Medical Center will be included.

Inclusion criteria: age > 18 years, able to sign the consent form, stable kidney function.

Exclusion criteria: end stage renal disease, acute kidney injury or need of dialysis three months prior the procedure, acute infection, acute inflammation, BMI > 40, malignancy and pregnancy.

The diagnosis of AKI will be made based on Kidney Disease Improving Global Outcomes (KDIGO) Clinical Practice Guideline 2012, by comparing the baseline and post-operative serum creatinine and cystatin C and monitoring urine output during the procedure and after the procedure for 24 hours.

Data Analysis: Results will be presented as mean ± standard deviation for quantitative data. A p value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years, able to sign the consent form, stable kidney function.

Exclusion Criteria:

* end stage renal disease
* acute kidney injury or need of dialysis three months prior the procedure
* acute infection
* acute inflammation
* malignancy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A single center prospective observational cohort study will be conducted. 100 patients undergoing elective laparoscopic cholecystectomy in the Galilee Medical Center will be included.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of AKI following a laparoscopic cholecystectomy | Up to one week after the procedure
  kidney function, included estimated GFR and urinary markers will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: Undecided